CLINICAL TRIAL: NCT07099365
Title: A Randomised Controlled Cross-over Feasibility Trial of a Self-guided Smartphone App to Support Psychological Adjustment in Long-term Physical Conditions Compared to Usual Charity Support
Brief Title: Psychological Adjustment to Long-term (PAL) Physical Conditions: A Randomised Cross-over Feasibility Trial of a Self-guided App
Acronym: PAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Avegen Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 45014
Record Dates: First submitted 2025-07-25; First posted 2025-08-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-01

CONDITIONS: Depression, Anxiety; Chronic Disease
Keywords: anxiety; depression; psychological distress; chronic disease; cognitive behavioural therapy
MeSH Terms: conditions — Depression; Anxiety Disorders; Chronic Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Orbi + Usual Charity Support (UCS) (Experimental): Participants randomised to this condition receive access to a self-guided smartphone app (Orbi) based on cognitive behavioural therapy principles in addition to Usual Charity Support (Orbi + UCS) to support Psychological Adjustment in long-term physical conditions.
  Interventions: Device: Orbi
- Usual Charity Support (UCS) (No Intervention): Participants randomised to this condition access Usual Charity Support (UCS) for their long-term physical condition(s). Resources provided by the charities include supportive listening, online support groups, information resources and local community support groups.

INTERVENTIONS:
Device: Orbi — Orbi is adapted from COMPASS, a web-based cognitive behavioural therapy (CBT) intervention based on the Transdiagnostic Model of Adjustment in Long-Term (physical) Conditions Model. Orbi is made up of 13 topics, each exploring a different challenge faced by individuals with a LTC(s). Orbi is a self-guided CBT programme with no therapist involvement.
  Arms: Orbi + Usual Charity Support (UCS)

SUMMARY:
This study is a two-arm, randomised controlled cross-over feasibility study with a nested, optional qualitative study. The intervention consists of a self-guided smartphone app (Orbi) based on cognitive behavioural therapy (CBT) principles, which is designed to support psychological adjustment in long-term physical conditions. Orbi is an app adaption of an existing, evidence-based web-based intervention COMPASS. The control condition consists of usual charity support (UCS) for the relevant long-term physical health conditions (LTCs). All charity support includes a helpline which can be accessed via telephone or email.

The goal of this trial is to evaluate the feasibility of Orbi and the main questions it aims to answer are:

1. Is Orbi a feasible and acceptable intervention for individuals experiencing psychological distress related to LTCs?
2. Which aspects of the Orbi app and the trial enhance or diminish participants' experiences?

Participants will:

* Be randomised and each participant has an equal (50 %) chance of being assigned either to the Orbi+UCS group or to UCS group alone for 12 weeks. After 12 weeks, they will be crossed over to the alternate condition for another 12 weeks
* Complete questionnaires to assess psychological distress and intervention engagement at baseline, 6 weeks, and 12 weeks.
* A subset of participants will be invited to take part in a nested, optional semi-structured interviews to explore their experiences using Orbi and participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18-years
* Verbal and written proficiency in English
* United Kingdom resident (General Practitioner registered)
* Basic computer literacy
* Email address to register with Orbi
* Have a long-term physical health condition
* Are experiencing distress related to their long-term physical condition

Exclusion Criteria:

* Evidence of substance dependency, cognitive impairment, severe mental health conditions identified by adhering to usual care Improving Access to Psychological Therapies (IAPT) screening practices that are employed at assessment and triage
* Those with evidence of severe depression and/ or anxiety scoring over 6 on the Patient Health Questionnaire-4 (PHQ-4) eligibility questionnaire or scoring 1 or above on the eligibility Patient Health Questionnaire-9 (PHQ-9) suicide risk question
* Receiving active psychological treatment from psychologist/counsellor/therapist or online psychological intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment | At baseline
  Frequencies and percentages of the number of potential participants recruited to the study
Retention | At baseline, 6 weeks (mid-study) and 12 weeks (end of study)
  Frequencies and percentages of the number of participants retained in the study
Reach | At baseline
  Frequencies and percentages of recruited participants who are from under-represented ethnic groups for research conducted in the United Kingdom (e.g. ethnic groups other than white British)
Acceptability | 6 weeks (mid-study) and 12 weeks (end of study)
  Quantitative: Frequencies and percentages or means and standard deviations of the Theoretical Framework of Acceptability (TFA) questionnaire
  Qualitative: Framework Thematic Analysis

SECONDARY OUTCOMES:
App usability | 6 weeks (mid-study) and 12 weeks (end of study)
  Qualitative: Usability of the app will be evaluated within the interviews and Framework Thematic Analysis.
Primary adherence and engagement: App usage data | 6 weeks (mid-study) and 12 weeks (end of study)
  Frequencies and percentages or means and standard deviations of:
  Number of intervention sessions accessed and/or completed; time spent or time to completion, number of log-ins, pages viewed.
Compare post intervention scores on Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS-15) adjusting for baseline differences between groups | At baseline, 6 weeks (mid-study) and 12 weeks (end of study)
  A 15-item scale assessing symptoms of anxiety and depression. It includes items from the Patient Health Questionnaire Scale (PHQ-8) for depression and the Generalised Anxiety Disorder Scale (GAD-7) for anxiety, each scored on a 4-point Likert scale from 'not at all' (0) to 'nearly every day' (3). Total scores range from 0 to 45 with higher scores indicating greater symptom severity.
Compare post intervention scores on Patient Health Questionnaire Scale - (PHQ-8) adjusting for baseline differences between groups | At baseline, 6 weeks (mid-study) and 12 weeks (end of study)
  8-item questionnaire scoring the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for depression on 4-point Likert scales from 'not at all' (0) to 'nearly every day' (3). Total scores below 5, 10, 15, 20, and up to 24 are categorised as none-to-minimal, mild, moderate, moderately severe, and severe depression.
Compare post intervention scores on Generalised Anxiety Disorder Scale (GAD-7) adjusting for baseline differences between groups | At baseline, 6 weeks (mid-study) and 12 weeks (end of study)
  A 7-item questionnaire assessing the severity of generalised anxiety symptoms based on DSM-IV criteria. Each item is scored on a 4-point Likert scale from 'not at all' (0) to 'nearly every day' (3). Total scores range from 0 to 21, with cut-off points at 5, 10, and 15, indicating mild, moderate, and severe anxiety, respectively.
Compare post intervention scores on Illness Related Distress (IRD) scale adjusting for baseline differences between groups | At baseline, 6 weeks (mid-study) and 12 weeks (end of study)
  A 14-item scale assessing how a long-term physical health condition has affected the psychological distress experienced by an individual over the last two weeks. Intrapersonal IRD = items 1-7 (cut-off = 15); Interpersonal IRD = items 8-14 (cut-off = 12).
  The scale is augmented by 3 additional items. Two horizontal visual analogue scales ranging from 0 to 10: One indicating the amount of psychological distress that is attributed to having one or more physical Long Term Condition (LTC) over the last two weeks; one indicating the severity of psychological distress related to the LTC over the last two weeks. The final item asks the respondent to specify which LTC they are attributing their psychological distress to (as many people are affected by multiple LTCs in parallel).
Compare post intervention scores on Work and Social Adjustment Scale (WSAS) adjusting for baseline differences between groups | At baseline, 6 weeks (mid-study) and 12 weeks (end of study)
  A 5-item scale measuring the impact of mental health issues on daily functioning across work, home management, social leisure, private leisure, and close relationships. Each item is scored from 0 (no impairment) to 8 (severe impairment). Total score ranges from 0 to 40, with higher scores indicating greater functional impairment.
Compare post intervention scores on EuroQol 5-Dimension 3-Level Questionnaire (EQ-5D-3L) adjusting for baseline differences between groups | At baseline, 6 weeks (mid-study) and 12 weeks (end of study)
  A 5-item scale measuring health-related quality of life across five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on three levels (1 to 3). Total score ranges from 5 to 15, with higher scores indicating more severe issues in health-related quality of life.
Compare post intervention scores on Patient Enablement Instrument (PEI) adjusting for baseline differences between groups | 6 weeks (mid-study) and 12 weeks (end of study)
  A 6-item questionnaire assessing patient enablement (i.e. patients' ability to understand and cope with their health and illness) on a 4-point scale (much better, better, same or less, not applicable). Total scores range from 0 to 12, with higher scores indicating greater patient enablement.
Compare post intervention scores on Patient Global Impression of Severity (PGI-S) adjusting for baseline differences between groups | At baseline, 6 weeks (mid-study) and 12 weeks (end of study)
  A one-item questionnaire assessing perceived severity of participants' long-term physical conditions using a 4-point scale with scoring ranges from 0 to 3. Higher scores indicate greater severity.
Compare post intervention scores on Patient Global Impression of Improvement (PGI-I) adjusting for baseline differences between groups | 6 weeks (mid-study) and 12 weeks (end of study)
  A one-item questionnaire assessing how patient's health condition has changed since the beginning of the study on a 7-point scale with scoring ranges from 0 to 6. Higher scores indicate greater deterioration.
Comparison between intervention and control groups on Health Service Utilisation | At baseline, 6 weeks (mid-study) and 12 weeks (end of study)
  Usage of health services will be captured with the Health Service Use Questionnaire. Participants will indicate whether they have accessed key services, including general practitioner (GP), psychological or counselling services, and emergency care during the past 3 months. For each service reported, additional items capture (i) the number of contacts, (ii) the mode of contact (e.g., in-person, telephone, video), and (iii) the duration of the most recent contact.
Comparison between intervention and control in access of charity services | 6 weeks (mid-study) and 12 weeks (end of study)
  Participants will also be asked about their access of charity resources. A multiple-selection drop-down box will show the following options (charity helpline, online forums/networks/phone counselling, information booklets, others)

CONTACTS AND LOCATIONS:
Overall Officials: Rona Moss-Morris, PhD, Principal Investigator — King's College London
Locations (1):
- Health Psychology Department, King's College London, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available on request from the corresponding author. The data will not be available publicly due to privacy or ethical restrictions.
Supporting Information: CSR
Access Criteria: The data will only be available on request.

REFERENCES:
- [Background] Carroll S, Moon Z, Hudson J, Hulme K, Moss-Morris R. An Evidence-Based Theory of Psychological Adjustment to Long-Term Physical Health Conditions: Applications in Clinical Practice. Psychosom Med. 2022 Jun 1;84(5):547-559. doi: 10.1097/PSY.0000000000001076. Epub 2022 Apr 12. PMID 35412516
- [Background] Hulme K, Hudson JL, Picariello F, Seaton N, Norton S, Wroe A, Moss-Morris R. Clinical efficacy of COMPASS, a digital cognitive-behavioural therapy programme for treating anxiety and depression in patients with long-term physical health conditions: a protocol for randomised controlled trial. BMJ Open. 2021 Oct 25;11(10):e053971. doi: 10.1136/bmjopen-2021-053971. PMID 34697123
- [Background] Picariello F, Hulme K, Seaton N, Hudson JL, Norton S, Wroe A, Moss-Morris R. A randomized controlled trial of a digital cognitive-behavioral therapy program (COMPASS) for managing depression and anxiety related to living with a long-term physical health condition. Psychol Med. 2024 Jun;54(8):1796-1809. doi: 10.1017/S0033291723003756. Epub 2024 Feb 14. PMID 38350600
- [Background] Seaton N, Moss-Morris R, Hulme K, Macaulay H, Hudson J. A cognitive-behavioural therapy programme for managing depression and anxiety in long-term physical health conditions: mixed-methods real-world evaluation of the COMPASS programme. BJPsych Open. 2023 Aug 11;9(5):e153. doi: 10.1192/bjo.2023.519. PMID 37563762